CLINICAL TRIAL: NCT06830603
Title: A Post Market, Prospective Clinical Study Evaluating Clinical and Radiographic Outcomes of Patients Undergoing Total Knee Arthroplasty with Physica TT Tibial Plate
Brief Title: Physica TT Tibial Plate Prospective Study
Status: Not yet recruiting | Type: Observational
Sponsor: Limacorporate S.p.a (Industry)
Responsible Party: Sponsor
Other Study IDs: K-41
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Knee Arthroplasty, Total; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Physica TT Tibial Plate: Total knee arthroplasty with Physica TT Tibial Plate

SUMMARY:
This prospective clinical study aims at evaluating clinical, radiographic, patient-reported outcomes of total knee arthroplasty with Physica TT Tibial Plate over 2 years after surgery, in order to assess the performance and safety of the devices. Short-term survivorship of the implant and the incidence of early complications are evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Patient requiring a total knee arthroplasty (TKA) and suitable for receiving Physica TT Tibial Plate;
2. Age ≥ 18 years old;
3. Candidate for primary total knee replacement when clinical indications based on physical examination and medical history include one or more of the following conditions:

   1. Non-inflammatory degenerative joint disease such as knee osteoarthritis, post traumatic knee arthritis;
   2. Inflammatory degenerative joint disease such as rheumatoid arthritis;
4. Patient has well-preserved and well-functioning collateral ligaments
5. Patient is able to understand the conditions of the study, is willing and able to follow all prescribed rehabilitation as well as willing to perform all scheduled follow-up visits;
6. Patient has signed the study-specific Informed Consent Form prior to study activities

Exclusion Criteria:

1. Patient is affected by one or more of the conditions that are stated as Physica contraindications for use, which are:

   * Severe instability of the knee joint secondary to the absence of collateral ligament integrity and/or function.
   * Any active or suspected infection (local or systemic) or previous history of infection that may affect the prosthetic joint.
   * Significant bone loss on femoral or tibial joint side.
   * Known incompatibility or allergy to the product materials, and/or metal hypersensitivity to implant materials.
   * Septicaemia.
   * Persistent acute or chronic osteomyelitis.
   * Open epiphyses (immature patient with active bone growth).
   * Necrotic bone
   * Arterial vascular insufficiency or nerve diseases of the lower limbs severe enough to interfere with the study evaluation.
   * Compromised bone stock due to disease, infection or prior implantation that cannot provide adequate support and/or fixation to the prosthesis.
   * Systemic or metabolic disorders leading to progressive bone deterioration, which may impair fixation and stability of the implant.
   * Any concomitant disease and dependency that might affect the performance of the implanted prosthesis.
   * Important osteoporosis, haemophilic disease.
   * Internistic problems with high risk for surgery.
2. Previous partial knee replacement (unicompartmental, bicompartmental or patellofemoral joint replacement), patellectomy, high tibial osteotomy.
3. Affected by malignant cancer with life expectancy less than 2 years or where cancer treatment might affect the normal postoperative course.
4. Any clinically major pathology based on clinical medical history or any medical intervention or reason that the Investigator feels may affect the study evaluation.
5. Neurological or musculoskeletal disorder or disease that may adversely affect gait, functional recovery and evaluation.
6. Neuromuscular or neurosensory deficit that would hamper the performance assessment of the device.
7. Any psychiatric illness that would prevent comprehension of the details and nature of the study.
8. Simultaneously taking part in another surgical intervention study or pain management study that may affect with clinical study outcomes.
9. Female patient who is pregnant, nursing, or planning a pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General population of subjects requiring a primary TKR with a diagnosis of painful primary or secondary osteoartrithis not responding to other conservative treatments, after the review of medical history and the radiographic evaluation of the affected knee.
Sampling Method: Non-Probability Sample
Enrollment: 142 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in Knee Society Score from preoperative to 2 years after surgery | From preoperative to 2 years after surgery
  0-100 scale. Scores rating from 80 to 100 are considered excellent, between 70 and 79 good, between 60 and 69 fair, and less than 60 poor

SECONDARY OUTCOMES:
Change in Oxford Knee Score | From preoperative to 2 years after surgery
  Overall score from 0 to 48, with 48 being the best outcome
Change in Range of Motion | From preoperative to 2 years after surgery
Radiographic implant evaluation and stability assessment | From preoperative to 2 years after surgery
  The treated knee is analyzed postoperatively based on knee x-rays. The following parameters are evaluated: - Presence of radiolucent lines - Presence of osteolysis - Presence of loosening - Presence of heterotopic ossification - Presence of periprosthetic fractures
Incidence, type and severity of Adverse Device Effects (ADE) and Serious Adverse Device Effects (SADE) | From preoperative to 2 years after surgery
Implant survival rate | From preoperative to 2 years after surgery